CLINICAL TRIAL: NCT04899141
Title: Prospective Registry of ihtDEStiny® Coronary Stent in Regular PCI Practice
Acronym: VELAZQUEZ
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC26-VELAZQUEZ
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
Keywords: Percutaneous Coronary Intervention; Drug Eluting Stent
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease
  Interventions: Device: Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Percutaneous Coronary Intervention — stenting with the ihtDEStiny® sirolimus eluting stent

SUMMARY:
Prospective registry intended to evaluate clinical outcomes of ihtDEStiny drug eluting coronary stent.

DETAILED DESCRIPTION:
Prospective registry intended to evaluate clinical outcomes of ihtDEStiny drug eluting coronary stent use in real-world percutaneous coronary intervention

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* PCI and stent implantation indication according to ESC Myocardial Revascularization Guidelines
* 1 or more stenosis at native coronary anatomy, in a 2-4mm vessel size, where 1 or more ihtDEStiny® drug eluting stent were implanted (or attempted to be implanted).
* Informed consent signed after PCI

Exclusion Criteria:

* Patient refusal to participate in the study
* Pregnancy
* Other DES implantation during index PCI, or 30 days before of after index PCI
* PCI at surgical grafts
* PCI for in-stent restenosis
* Killip class 3-4 Acute Coronary Syndromes (ACS)
* High bleeding risk with dual antiplatelet intolerance for at least 3 months (or 6 months for ACS PCI)
* Allergy or hypersensitivity to sirolimus
* Patients requiring surgery (cardiac or non-cardiac) in the next 3 months after index PCI
* Patients with life expectancy <2 years
* Patients included in other trials or clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with all inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 2 years
  Rate of target lesion failure
Death | 2 years
  Death
Target vessel myocardial infarction | 2 years
  Target vessel myocardial infarction
Target lesion revascularization (TLR) | 2 years
  Target lesion revascularization (TLR)
Cardiovascular Death | 2 years
  Cardiovascular Death

SECONDARY OUTCOMES:
Stent thrombosis | 2 years
  Stent thrombosis
Target Vessel Failure (TVF) | 2 years
  Composite event of cardiovascular (CV) death, target vessel myocardial infarction (MI) and target vessel revascularization (TVR)
Major Adverse Cardiovascular Event (MACE) | 2 years
  Composite event of cardiovascular (CV) death, non-fatal myocardial infarction (MI) and non-fatal stroke
Patient Oriented Composite Event | 2 years
  Composite event of death, non-fatal myocardial infarction (MI), non-fatal stroke or any revascularization
Severe BARC Bleeding | 2 years
  BARC Bleeding ≥3
Device success | During procedure
  residual coronary stenosis<50%, normal coronary flow and absence of coronary dissection ≥C
Procedural success | 3 days
  Device success and absence of PCI complication (periprocedural MI, coronary perforation, urgent CABG or death) or revascularization within 3 days

CONTACTS AND LOCATIONS:
Locations (20):
- Centro Hospitalar Universitario Do Algarbe, Faro, Portugal
- Spain (19):
  - Hospital Universitario Regional de Malaga Carlos Haya, Málaga, Malaga
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital General Universitario de Elche, Elche
  - Hospital de Galdakao, Galdakao
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Lucus Agusti, Lugo
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital Universitario Virgen Arrixaca, Murcia
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario de Araba, Vitoria-Gasteiz
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] de la Torre Hernandez JM, Ocaranza Sanchez R, Santas Alvarez M, Pinar Bermudez E, Hurtado Martinez JA, Garcia Del Blanco B, Otaegui I, Fernandez Nofrerias E, Carrillo Suarez X, Sainz Laso F, Casanova Sandoval JM, Rivera Aguilar PK, Cid B, Trillo R, Lozano Ruiz-Poveda F, Peral Disdier V, Telleria M, Torres A, Sanchis J, Oliva X, Freixa X, Sadaba Sagredo M, Moreu J, Hernandez F. Comparison of One-Year Outcomes Between the ihtDEStiny BD Stent and the Durable-Polymer Everolimus- and Zotarolimus-Eluting Stents: A Propensity-Score-Matched Analysis. Cardiovasc Revasc Med. 2021 Oct;31:1-6. doi: 10.1016/j.carrev.2020.09.046. Epub 2020 Oct 3. PMID 33060037
- [Background] de la Torre Hernandez JM, Otaegui I, Subinas A, Gomez-Menchero A, Moreno R, Rondan J, Munoz-Garcia E, Sainz-Laso F, Garcia Del Blanco B, Rumoroso JR, Diaz JF, Berenguer A, Gomez-Lara J, Zueco J. First-in-Man Evaluation of a Sirolimus-Eluting Stent With Abluminal Fluoropolymeric/Triflusal Coating With Ultrathin Struts by OCT at 9 Months' Follow-Up: The PROMETHEUS Study. Cardiovasc Revasc Med. 2021 Nov;32:18-24. doi: 10.1016/j.carrev.2020.12.025. Epub 2020 Dec 29. PMID 33386256
- [Background] Buiten RA, Ploumen EH, Zocca P, Doggen CJM, Danse PW, Schotborgh CE, Scholte M, van Houwelingen KG, Stoel MG, Hartmann M, Tjon Joe Gin RM, Somi S, Linssen GCM, Kok MM, von Birgelen C. Thin, Very Thin, or Ultrathin Strut Biodegradable or Durable Polymer-Coated Drug-Eluting Stents: 3-Year Outcomes of BIO-RESORT. JACC Cardiovasc Interv. 2019 Sep 9;12(17):1650-1660. doi: 10.1016/j.jcin.2019.04.054. Epub 2019 Aug 14. PMID 31422087
- [Background] El-Hayek G, Bangalore S, Casso Dominguez A, Devireddy C, Jaber W, Kumar G, Mavromatis K, Tamis-Holland J, Samady H. Meta-Analysis of Randomized Clinical Trials Comparing Biodegradable Polymer Drug-Eluting Stent to Second-Generation Durable Polymer Drug-Eluting Stents. JACC Cardiovasc Interv. 2017 Mar 13;10(5):462-473. doi: 10.1016/j.jcin.2016.12.002. PMID 28279314
- [Background] Iantorno M, Lipinski MJ, Garcia-Garcia HM, Forrestal BJ, Rogers T, Gajanana D, Buchanan KD, Torguson R, Weintraub WS, Waksman R. Meta-Analysis of the Impact of Strut Thickness on Outcomes in Patients With Drug-Eluting Stents in a Coronary Artery. Am J Cardiol. 2018 Nov 15;122(10):1652-1660. doi: 10.1016/j.amjcard.2018.07.040. Epub 2018 Sep 8. PMID 30292330